CLINICAL TRIAL: NCT06219291
Title: Preventing the Progression of Physical Disability and Promoting Brain Functional Adaptation in People With Multiple Sclerosis: Integration of Early Rehabilitative Treatment and Multimodal Clinical and Instrumental Assessment - Part A
Brief Title: Preventing the Progression of Multiple Sclerosis: Early Rehabilitative Treatment and Multimodal Assessment - Part A
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: IRCCS San Raffaele (Other); Azienda Sanitaria Locale di Cagliari (Other)
Responsible Party: Sponsor
Other Study IDs: 03_17/02/2021 Part A
Record Dates: First submitted 2023-09-11; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: early phase; non-disabled
MeSH Terms: conditions — Multiple Sclerosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observation of the natural course of the disease

SUMMARY:
Motor performance of people with Multiple Sclerosis (PwMS) can decline since the onset of the disease.

Longitudinal studies are needed to detect early worsening in mobility and balance using wearable devices for activity tracking and neurophysiological techniques for investigating brain functional adaptation. Similarly, neurophysiological assessment can provide evidences on the integrity of brain motor networks and mechanisms underlying cortical plasticity in the early disease phase, potentially providing a set of reliable prognostic factors of disease progression in early diagnosed PwMS.

Furthermore, disease progression might be delayed using physical activity, which is effective in PwMS with moderate disability to ameliorate mobility and promoting brain reorganization and seems promising also for PwMS in the early stages of the disease. Functional Near-Infrared Spectroscopy (fNIRS) measures blood flow which accompanies neuronal activity, thus, it can provide spatial information about changes in cortical activation patterns and it could represent a useful tool for studying the effect of exercise on cortical plasticity. The aims of the study in non-disabled PwMS are: 1) a) to assess the presence of subclinical balance and walking impairments using wearable devices and multimodal gait analysis and b) to investigate cortical activity during exercise, 2) to define prognostic factors associated to disease progression and 3) to study the efficacy of physical activity in preventing the worsening of mobility and stimulating brain functional adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Stable disease course (without worsening over 1 point at the EDSS in the last 3 months)
* Expanded Disability Status Scale (EDSS) <2.5

Exclusion Criteria:

* Major depression
* Mini-Mental State Examination < 27
* Other cardiovascular or orthopedic diseases that interfere with physical exercise
* Undefined or not confirmed diagnosis of MS (Polman criteria)
* Progressive course of the disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited within Persons with Multiple Sclerosis attending the clinical centers for routine medical visits willing to participate to the study after the presentation of the information sheet.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk test (SMWT) | Baseline, Follow-up 1year, Follow-up 2year
  Assesses distance in meters walked over 6 minutes as a sub-maximal test of endurance capacity.

SECONDARY OUTCOMES:
Concentration of oxygenated hemoglobin (Delta oxyHb) | Baseline, Follow-up 1year, Follow-up 2year
  The differences in oxyHb during task period and resting state. Data will be extracted from functional Near InfraRed Spectroscopy (fNIRS) assessment.
Expanded Disability Status Scale (EDSS) | Baseline, Follow up 1year, Follow up 2year
  Assess the neurological impairment as a result of Multiple Sclerosis, ranging from 0 (normal neurological exam) to 10 (death due to Multiple Sclerosis).
Regularity of gait | Baseline, Follow-up 1year, Follow-up 2yearr
  Instrumental gait indexes will be extracted from an Inertial Measurement Unit (IMU) during the a walking test.

OTHER OUTCOMES:
Dual Task Cost | Baseline, Follow-up 1year, Follow-up 2year
  The physical and mental cost of the contemporary execution of two tasks will be evaluated with a specific test (walking and counting backwards). The dual-task cost quantifies this interference and is the percentage change of dual-task (DT) performance compared with single-task performance.
  Moreover, we will assess the patients' perspective on the perceived difficulties of dual-tasking during daily activities through the Dual-task Impact on Daily-living Activities Questionnaire (DIDA-Q). The questionnaire is composed by 19 items. It provides a global score ranging on a 0-76 scale and three subscale scores identifying the components mostly contributing to the perceived difficulty in DT activities: balance and mobility (6 items, score range 0-24), cognition (8 items, score range 0-32) and upper-limb ability (5 items, score range 0-20). Higher scores represent greater difficulties in performing dual task activities.
Dual-task Impact on Daily-living Activities Questionnaire (DIDA-Q) | Baseline, Follow-up 1year, Follow-up 2year
  Investigators will assess the patients' perspective on the perceived difficulties of dual-tasking during daily activities through the Dual-task Impact on Daily-living Activities Questionnaire (DIDA-Q). The questionnaire is composed by 19 items. It provides a global score ranging on a 0-76 scale and three subscale scores identifying the components mostly contributing to the perceived difficulty in DT activities: balance and mobility (6 items, score range 0-24), cognition (8 items, score range 0-32) and upper-limb ability (5 items, score range 0-20). Higher scores represent greater difficulties in performing dual task activities.
Timed 25 foot walk (T25FWT) | Baseline, Follow-up 1year, Follow-up 2year
  Evaluation of gait velocity (m/s) derived from the time taken to cover a distance of 25 foot.
Fullerton Advanced Balance Scale - Short version (FAB-s) | Baseline, Follow-up 1year, Follow-up 2year
  A test to evaluate static and dynamic balance composed by 8 tasks. Each task is rated from 0 (impossible) to 4 (normal execution). Higher values represent better balance capacity.
Explosive power | Baseline, Follow-up 1year, Follow-up 2year
  To evaluate explosive power capacity, subjects will execute bipodalic squat and counter-movement jumps (mono e bipodalic) wearing an IMU (g-Walk, BTS). Data regarding jump height, power, velocity and force will be extracted through the dedicated software (Baiobit, BTS).
Tactile sensitivity (Monofilament Test) | Baseline, Follow-up 1year, Follow-up 2year
  Monofilament test will be applied to the eminence of the distal phalanx of the hallux to test levels of touch sensitivity of the foot. The patient close his eyes and say "yes" every time touch is felt. The level of sensitivity is determined by the smallest monofilament felt correctly for three times. Level of sensitivity thus will be classified from loss of deep protective sensation to normal light touch.
Nine Hole peg Test (NHPT) | Baseline, Follow-up 1year, Follow-up 2year
  A measure to assess fine dexterity.Is administered by asking the client to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container. Scores are based on the time taken to complete the activity, recorded in seconds. Normal scores are around 18 seconds.
The revised Brief Visuospatial Memory Test (BVMTR): | Baseline, Follow-up 1year, Follow-up 2year
  Is a measure of visual memory ability. Six abstract designs are presented for 10 sec and patients render the stimuli. Each design receives from 0 to 2 points representing accuracy and location. The test is repeated 3 times and the final scores is the sum of the three trials.
California Verbal Learning Test (CVLT2): | Baseline, Follow-up 1year, Follow-up 2year
  It measures verbal memory ability. Patients listen to a 16 list of word and report as many of the items as possible. There are five learning trials. The total score is the total number of recalled items over the five learning trials.
Symbol Digit Modalities Test (SDMT) | Baseline, Follow-up 1year, Follow-up 2year
  It assesses mental processing speed. It presents a series of nine symbols, paired with a single digit. Patients are asked to voice the digit associated with each symbol for 90 sec. The scores is the number correct over the 90 sec time span.
Multiple Sclerosis Walking Scale 12 (MSWS-12) | Baseline, Follow-up 1year, Follow-up 2year
  Is a self-report measure of the impact of Multiple Sclerosis on the individual's walking ability. The scoring provides options 1-5 for each item, with 1 meaning no limitation and 5 meaning extreme limitation on the gait-related item.
Fatigue Severity Scale (FSS) | Baseline, Follow-up 1year, Follow-up 2year
  Is a 9-item self-administered questionnaire to measure the perceived impact of fatigue. The minimum score is 9 and maximum score possible is 63. Higher scores represent greater fatigue severity. If the score is calculated as the mean score of the 9 items, the cut-off score for the presence of the symptom fatigue is set as scores higher than 4.
Community Integration Questionnaire (CIQ) | Baseline, Follow-up 1year, Follow-up 2year
  Is a self-administered questionnaire used to assess the social role limitations and community interactions. Score ranges from 0 (no integration) to 29 (full participation).
Hospital Anxiety and Depression Scale (HADS) | Baseline, Follow-up 1year, Follow-up 2year
  A questionnaire to detect the presence of anxiety and depression. Subscores are calculated for anxiety and depression ranging from 0 (normal) to 21 (abnormal) with a cut-off score of 8.
Lifetime Total Physical Activity Questionnaire (LTPAQ) | Baseline, Follow-up 1year, Follow-up 2year
  is an interviewer-administered questionnaire used to estimate a respondent's physical activity done from childhood to the present in terms of months, days and hours. Data will be compared to normative values collected from a comparable sample of healthy subjects.
Amount of physical activity | Baseline, Follow-up 1year, Follow-up 2year
  Subjects will be monitored for 1 week wearing an actigraph (GENEActiv). Actigraphy is a non-invasive method of monitoring human rest/activity cycles through a wereable accelerometer. Data for rest/active period will be extracted through a dedicated software.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Rovaris, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi; Raffaella Chieffo, MD, Principal Investigator — IRCCS Ospedale San Raffaele; Eleonora Cocco, MD, Principal Investigator — Ospedale Binaghi ASL Cagliari, Sardegna
Locations (3):
- Italy (3):
  - Ospedale Binaghi ASL Cagliari, Cagliari
  - IRCCS Ospedale San Raffele, Milan
  - IRCCS Fondazione Don Carlo Gnocchi, Milan

REFERENCES:
- [Derived] Gervasoni E, Torchio A, Bertoni R, Chieffo R, Rocca MA, Pau M, Cocco E, Morozumi T, Filippi M, Cattaneo D, Rovaris M. Beyond EDSS: multidomain impairments are detectable and associated with walking disorders in low-disabled people with multiple sclerosis. J Neurol. 2025 May 18;272(6):404. doi: 10.1007/s00415-025-13128-7. PMID 40382461